CLINICAL TRIAL: NCT06314893
Title: Correlation of High Resolution Manometry and Upper Gastrointestinal Marshmallow Study in Preoperative Esophageal Motility Assessment
Brief Title: Establishing a Correlation Between HRM and UGI MM Studies
Acronym: MMvsMANO
Status: Terminated | Type: Observational
Why Stopped: Study design revision
Sponsor: Lexington Health Incorporated (Other)
Responsible Party: Principal Investigator, Marc Antonetti, MD, Principal Investigator, Lexington Health Incorporated
Other Study IDs: LMCII2022-001
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Motility Disorders
Keywords: GI tract
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A retrospective and prospective cohort, quantitative data collection with the goal of comparing preoperative High Resolution Manometry HRM results to Upper Gastrointestinal Marshmallow ,UGI MM results, in patients undergoing preoperative esophageal motility assessments. The aim of this study is to establish a correlation between HRM and UGI MM in order to create a clinically supported gold standard measurement for preoperative esophageal motility assessment.

DETAILED DESCRIPTION:
Identifying esophageal motility disorders prior to surgical intervention is imperative when determining the procedural route that will produce the greatest positive patient outcome and reduce postoperative sequelae related to preoperative conditions. Possible disparities have been identified between HRM and UGI MM assessment results. Identifying testing variables and standards that could impact the obtained results will allow providers the ability to create a more customized plan of care and increase outcome predictability. Therefore, examining HRM and UGI MM level of agreement is essential to providing the best evidence-based practice care and meeting the unique needs of individual patients.

Currently, HRM results are noted as the standard benchmark for adequate assessment of esophageal motility function and disorders. Esophageal manometry testing provides a means to determine if the esophagus is functioning properly through a series of wet swallows. As a patient swallows, the esophagus contracts in a orderly sequence to push the swallowed contents to the stomach. Once the contents enter the stomach, the Lower Esophageal Sphincter, LES closes to prevent backflow or reflux of the stomach contents into the esophagus. Assessment of motility and sphincter function is vital prior to any surgical intervention that involves manipulation of the gastroesophageal junction,GEJ or surrounding structures. Inaccurate surgical manipulation can cause undesired pressure changes and alterations in normal peristalsis within the esophageal body. Any impairment to esophageal motility can compromise clearance and sphincter function, leading to adverse outcomes such as the development of intestinal metaplasia due to prolonged exposure of the mucosa to gastric acid

1.Patient Identification

1. Patients undergoing esophageal motility evaluation prior to surgical intervention. Surgical interventions involve manipulation of the upper gastrointestinal tract and immediate surrounding structures.
2. Patients undergoing procedures where the standard of care routinely includes preoperative motility assessment. These procedures include fundoplication procedures, open, laparoscopic and endoscopic and gastric sleeve or bypass candidates.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative patients who have undergone both HRM and UGI MM assessments as part of their preoperative plan of care.
2. Patients who have had surgical procedures involving the upper GI tract and immediate surrounding structures after completing HRM and UGI MM assessments preoperatively
3. Adults age 18 and older

Exclusion Criteria:

1. Patients who continued taking narcotics, calcium channel blockers, nitrates or promotility medications the day of the HRM test, as these medications could falsely relax or hyper stimulate esophageal structures.
2. Patients with a past surgical history that includes Heller myotomy, peroralesophageal myotomy, botulinum injections, pneumatic dilations or gastric fundoplication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing preoperative testing for surgical intervention involving manipulation of the upper gastrointestinal tract.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Determining the correlation between HRM and UGI MM assessments among preoperative candidates will provide an evidenced based evaluation strategy for establishing procedural candidacy and predicting postoperative outcomes. | June 2021 -July 2025

CONTACTS AND LOCATIONS:
Overall Officials: Marc Antonetti, MD, Principal Investigator — Lexington Health Incorporated
Locations (1):
- Lexington Health Incorporated, West Columbia, South Carolina, United States

REFERENCES:
- [Background] Yadlapati R. High-resolution esophageal manometry: interpretation in clinical practice. Curr Opin Gastroenterol. 2017 Jul;33(4):301-309. doi: 10.1097/MOG.0000000000000369. PMID 28426462
- [Background] FalcAo AM, Nasi A, Szachnowicz S, Santa-Cruz F, Seguro FCBC, Sena BF, Duarte A, Sallum RA, Cecconello I. Does the nissen fundoplication procedure improve esophageal dysmotility in patients with barrett's esophagus? Rev Col Bras Cir. 2020 Nov 30;47:e20202637. doi: 10.1590/0100-6991e-20202637. eCollection 2020. English, Portuguese. PMID 33263652
- [Background] Musella M, Vitiello A, Berardi G, Velotti N, Pesce M, Sarnelli G. Evaluation of reflux following sleeve gastrectomy and one anastomosis gastric bypass: 1-year results from a randomized open-label controlled trial. Surg Endosc. 2021 Dec;35(12):6777-6785. doi: 10.1007/s00464-020-08182-3. Epub 2020 Dec 2. PMID 33269429
- See also: Esophageal Manometry — http://www.ncbi.nlm.nih.gov/books/NBK559237